CLINICAL TRIAL: NCT05980676
Title: Starting a Weekday Outdoor Walking (WOW) Routine: A Randomized Controlled Study
Brief Title: Starting a Weekday Outdoor Walking (WOW) Routine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-014
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Physical Inactivity
Keywords: Behavioral health; Health behavior change; Habit formation; Implementation intentions
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician performing statistical analysis will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group will be told that they can work a WOW routine on their own, with the opportunity to complete the intervention after completing the 4-week follow-up assessment.
- No-Coach (Experimental): This is a fully automated intervention. The No-Coach group will complete an online activity that will guide the creation of a habitual instigation implementation intention (e.g., When I finish eating lunch at work, then I will put on my walking shoes and go outside) and receive a 2-week long personalized email campaign. They will not be able to reply to the emails for support.
  Interventions: Behavioral: Personalized Two-Week Email-Based Program
- Coached (Experimental): This is a semi-automated intervention. The Coached group will complete an online activity that will guide the creation of a habitual instigation implementation intention (e.g., When I finish eating lunch at work, then I will put on my walking shoes and go outside) and receive a 2-week long personalized email campaign. Prompts will be added to the end of each email such that these participants can respond to give feedback, ask questions, and receive additional support from a (human) coach.
  Interventions: Behavioral: Personalized Two-Week Email-Based Program

INTERVENTIONS:
Behavioral: Personalized Two-Week Email-Based Program — Both intervention groups will complete an activity that will guide the creation of a habitual instigation implementation intention (e.g., When I finish eating lunch at work, then I will put on my walking shoes and go outside) and receive a 2-week long personalized email campaign. The Coached group will be able to reply to the emails to give feedback, ask questions, and receive additional support.
  Arms: Coached; No-Coach

SUMMARY:
The purpose of this 4-week randomized study is to evaluate the effect of personalized plans plus an email campaign, with and without email-based coaching (eCoaching), on engagement in a new weekday outdoor walking (WOW) routine and average daily step count. Approximately 150 participants will be recruited via paid ads on Facebook and Instagram. Participants will be randomized to a control group, an intervention group without eCoaching, and an intervention group with eCoaching. The control group will be told that they can work a WOW routine on their own, with the opportunity to take part in the intervention after completing the 4-week follow-up assessment. Both intervention groups will complete an activity that will guide the creation of habit plan (e.g., When I finish eating lunch at work, then I will put on my walking shoes and go outside) and receive a 2-week long personalized email campaign. The primary outcome of interest is change in average daily step count from the month prior to the month after baseline assessment, as compared across the three groups. It is hypothesized that the intervention groups will result in an increase in daily step count, as compared to the control group. Secondary outcomes include habit strength at one-month follow-up and change in self-reported sleep quality and self-efficacy from baseline to follow-up.

DETAILED DESCRIPTION:
The purpose of this 4-week randomized study is to evaluate the effect of personalized implementation intentions plus an email campaign, with and without email-based coaching (eCoaching), on engagement in a new weekday outdoor walking (WOW) routine and average daily step count. Approximately 150 participants will be recruited via paid ads on Facebook and Instagram. Participants will be randomized (1:1:1) to a control group, an intervention group without eCoaching, and an intervention group with eCoaching. The control group will be told that they can work a WOW routine on their own, with the opportunity to take part in the intervention after completing the 4-week follow-up assessment. Both intervention groups will complete an activity that will guide the creation of a habitual instigation implementation intention (e.g., When I finish eating lunch at work, then I will put on my walking shoes and go outside) and receive a 2-week long personalized email campaign. The primary outcome of interest is change in average daily step count from the month prior to the month after baseline assessment, as compared across the three groups. It is hypothesized that the intervention groups will result in a statistically significant increase in daily step count, as compared to the control group. Secondary outcomes include instigation habit strength (via Self-Report Behavioral Automaticity Index) at one-month follow-up and change in self-reported sleep quality (via the Single Items Sleep Quality Scale) and general self-efficacy (via General Self-Efficacy Scale) from baseline to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Indicates desire to increases daily step count
* Indicates having a safe and convenient location to conduct outdoor walks
* Uses an iPhone
* Can upload step count screenshots
* Intends to bring their phone on their walks
* Has email address that they check ~daily
* Has an average daily step count for month prior to enrolling <5,000/day, as determined by phone step data (screenshot submitted for verification).

Exclusion Criteria:

* Any medical issues that could be worsened by walking. This will be assessed via the Physical Activity Readiness Questionnaire (PAR-Q), minus the question asking the participant if they take medication for blood pressure or a heart condition. Researchers feel this question is overly cautious and would exclude many individuals who would otherwise qualify and benefit from walking regularly.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in average daily step count | Four weeks
  Change in average daily step count from the month prior to the month after baseline assessment, as compared across the three groups.

SECONDARY OUTCOMES:
Instigation habit strength | Four weeks
  Instigation habit strength measured via Self-Report Behavioral Automaticity Index at one-month follow-up. Scores range from 4-20, with a higher score indicating greater habit strength.
Change in sleep quality | Four weeks
  Change in self-reported sleep quality, measured via the Single Items Sleep Quality Scale, from baseline to follow-up. Scores range from 0=terrible sleep to 10=excellent sleep.
Change in general self-efficacy | Four weeks
  Change in general self-efficacy, measured via the New General Self-Efficacy Scale from baseline to follow-up. Scores range from 8-40, with a higher score indicating higher general self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Hollingsworth, PharmD, PhD, Principal Investigator — Assistant Professor at VCOM-Auburn
Locations (1):
- Edward Via College of Osteopathic Medicine-Auburn Campus (VCOM-Auburn), Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No